CLINICAL TRIAL: NCT03401008
Title: Descriptive Study of Buccodental Manifestations in a Group of Acromegalic Patients (AcroDent) Followed in the Endocrinology/Diabetology Service in the CHU of Clermont-Ferrand
Brief Title: Buccodental Manifestations in Patients With Acromegaly
Acronym: AcroDent
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-367
Record Dates: First submitted 2017-11-20; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Acromegaly
Keywords: Acromegaly; Oral manifestations
MeSH Terms: conditions — Acromegaly; Oral Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acromegalic patients: patients with a proven diagnosis of acromegaly achieved by an IGFA assay and a GH measure.
  Interventions: Other: Oral manifestations

INTERVENTIONS:
Other: Oral manifestations — To do the most accurate clinical and radiological state of oral manifestations in the series of prevalent acromegaly patients followed in the endocrinology service of the CHU of Clermont-Ferrand.

SUMMARY:
Context: Acromegaly is the rare condition (3 to 4 new cases per million per year) due to Growth Hormone (GH) overproduction by a somatotrope pituitary adenoma, resulting in Insulin Growth Factor 1 (IGF-1) excess. Consequently, many tissues of the organism become hypertrophied. Hypertrophy of gingival and dental tissues can lead to alteration of oral health. However, there are very few published data concerning oral impact of acromegaly.

Objective: To do the most accurate clinical and radiological state of oral manifestations in the series of prevalent acromegaly patients followed in the endocrinology service of the CHU of Clermont-Ferrand.

DETAILED DESCRIPTION:
Context/ study relevance: Acromegaly is a rare condition (3 to 4 new cases per million per year) due to Growth Hormone (GH) overproduction by a somatotrope pituitary adenoma, resulting in Insulin Growth Factor 1 (IGF-1) excess. Consequently, a dysmorphic syndrome prevailing at the level of face and extremities progressively develops associated with potentially severe general manifestations (cardiovascular, respiratory and metabolic complications). Oral manifestations of acromegaly are not well known, there is very few published data on this topic and a controversy about the existence of a parodontal disease, i.e. the presence of gingival sulcus deepening which can lead to tooth loss. IGF-1 excess could lead to gingival hypertrophy and then to gingival sulcus deepening. Otherwise, the dental cementum, the only dental tissue which can grow during all lifetime, could be influenced by an excess of IGF-1. It is likely that acromegaly is associated with pathological cementum hypertrophy.

Objective: To do the most accurate clinical and radiological state of oral manifestations in the series of prevalent acromegaly patients followed in the endocrinology service of the CHU of Clermont-Ferrand. Investigator will take a special interest in parodontal status i.e. the state of supporting tissues of the teeth and structural anomalies of dental cementum.

As secondary objective, investigator would make a histological characterization of gingival and dental (cementum) tissues when a surgical treatment of the oral condition is required. Investigator will search hypertrophic anomalies linked with GH/IGF-1 excess.

Material and methods: This is an observational, descriptive, cross-sectional, monocentric study conducted in the endocrinology/diabetology service of Clermont-Ferrand University Hospital (CHU), in France, where a series of about 70 prevalent acromegaly patients is annually followed. The participants will be adult acromegaly patients followed in this service, with proven diagnosis of acromegaly or previous acromegaly. They will be excluded of the study if they are totally toothless, if they take a medication associated with gingival hypertrophy if they are in a medical or chirurgical condition interacting with oral health so that the oral evaluation is not reliable or if there is no possibility of written informed consent. For each participant, investigator will collect demographic data and history of the pathology including previous and actual complications, biological tests results, imaging exams results and treatments. The participants will answer 3 questionnaires: AcroQol (quality of life in acromegaly patients), GOHAI (General Oral Health Assessment Index) and EPICES (evaluation of precariousness). The primary outcome will be a quantitative assessment of the oral health of the acromegalic patients with detailed assessment of 3 criteria:

* Depth of gingival sulcus measured for of all teeth
* CAO index (number of teeth with cavity or obturation or missing)
* Thickness of dental cementum on orthopantomogram and all other abnormality on this exam.

The secondary outcome will be the histological analysis of gingival and dental tissues if available.

All these measures will be taken during a routine odonto-stomatological consultation, part of the annual pathology evaluation at the endocrinology/diabetology service.

ELIGIBILITY:
Inclusion Criteria:

* Adult acromegal patient followed in the endocrinology/diabetology service of the CHU of Clermont-Ferrand
* Proven diagnosis of acromegaly or previous acromegaly

Exclusion Criteria:

* Minor subject
* Subject under guardianship or curatorship
* Total toothless patients
* No possibility of written informed consent
* Medical or chirurgical conditions interacting with oral health so that the oral evaluation is not reliable
* Medication associated with gingival hypertrophy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acromegalic patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
oral health of acromegal patients | at day 1 (during the odonto-stomatological consultation)
  the periodontal status would be determinate by measuring the depth of gingival sulcus with a graduated periodontal probe on the four dental faces (mesial, distal, vestibular and lingual), on each tooth present in the mouth.

SECONDARY OUTCOMES:
study of the dental cementum | at day 2 (24h after receipt of sample)
  the thickness of dental cementum would be measured on orthopantomogram. This characteristic could determinate the presence or not of hypercementosis
Determinate the CAO index | at day 2 (24h after receipt of sample)
  The CAO index could be determinate by counting the number of teeth with cavity or obturation or missing
Analysis of pathological gingival tissues | at day 2 (24h after receipt of sample)
  : if a gingival hypertrophy is determinate, a gingivectomy will be carried out and the tissue will be sent to the Anatomo-pathology laboratory to determinate its histological characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Igor TAUVERON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France